CLINICAL TRIAL: NCT02366195
Title: A Phase 2, Multicenter, Open-label, Single-arm Trial to Evaluate the Correlation Between Objective Response Rate and Baseline Intratumoral CD8+ Cell Density in Subjects With Unresected Stage IIIB to IVM1c Melanoma Treated With Talimogene Laherparepvec
Brief Title: Single-arm Trial to Evaluate the Role of the Immune Response to Talimogene Laherparepvec in Unresected Melanoma
Acronym: TVEC-325
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120325; 2013-005552-15 (EudraCT Number)
Record Dates: First submitted 2014-11-11; First posted 2015-02-19 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Unresected Stage IIIb to IVM1c Melanoma
Keywords: T-VEC; CD8+ cell density; objective response rate; unresected; Melanoma
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Talimogene Laherparepvec (Experimental): Talimogene laherparepvec was administered by intralesional injection into injectable cutaneous, subcutaneous, and nodal lesions at an initial dose of 10⁶ plaque-forming units (PFU) per mL on day 1 followed by a dose of 10⁸ PFU/mL 21 days after the initial dose and every 14 days thereafter. Participants were treated with talimogene laherparepvec until they achieved a complete response, all injectable tumors had disappeared, clinically significant (resulting in clinical deterioration or requiring change of therapy) disease progression beyond 6 months of treatment, per modified World Health Organization (WHO) response criteria, or intolerance of study treatment, whichever occurred first.
  Interventions: Drug: Talimogene Laherparepvec

INTERVENTIONS:
Drug: Talimogene Laherparepvec — The initial dose of talimogene laherparepvec is up to 4.0 mL of 10^6 PFU/mL. Subsequent doses of talimogene laherparepvec are up to 4.0 mL of 10^8 PFU/mL.
  Other Names: IMLYGIC®

SUMMARY:
The study is a phase 2, multi centered, single arm study designed to evaluate the correlation between cluster of differentiation 8-positive (CD8+) cell density and objective response rate in adults with unresected stage IIIB to IVM1c melanoma. This study will also evaluate the safety and tolerability profile of talimogene laherparepvec.

DETAILED DESCRIPTION:
The study will explore the hypothesis that intratumoral CD8+ cell density at baseline correlates with objective response rate in adults with unresected stage IIIB to IVMIc melanoma treated with talimogene laherparepvec.

ELIGIBILITY:
Inclusion Criteria:

1. Provided informed consent prior to initiation of any study-specific activities/procedures
2. Subject with stage IIIB to IVM1c melanoma for whom surgery is not recommended
3. Candidate for intralesional therapy
4. Measurable disease with greatest diameter ≥ 10 mm
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Adequate organ function

Other Inclusion Criteria May Apply

Exclusion Criteria:

1. Clinically active cerebral metastases.
2. Bone metastases
3. Primary ocular or mucosal melanoma
4. Active herpetic skin lesions or prior complications of herpes simplex virus type 1 (HSV-1) infection (eg, herpetic keratitis or encephalitis)
5. Requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (eg, acyclovir), other than intermittent topical use
6. Female subject is pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of talimogene laherparepvec
7. Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception

Other Exclusion Criteria May Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2020-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (38):
- Research Site, Salt Lake City, Utah, United States
- Austria (2):
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Liège
- France (5):
  - Research Site, Boulogne-Billancourt
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Poitiers
- Germany (4):
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Hanover
  - Research Site, Heidelberg
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion - Crete
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Pécs
  - Research Site, Szeged
- Italy (3):
  - Research Site, Bergamo
  - Research Site, Milan
  - Research Site, Siena
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Groningen
- Poland (2):
  - Research Site, Konin
  - Research Site, Warsaw
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Spain (5):
  - Research Site, Donostia / San Sebastian, Basque Country
  - Research Site, Badalona, Catalonia
  - Research Site, Barcelona, Catalonia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- United Kingdom (2):
  - Research Site, London
  - Research Site, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Malvehy J, Samoylenko I, Schadendorf D, Gutzmer R, Grob JJ, Sacco JJ, Gorski KS, Anderson A, Pickett CA, Liu K, Gogas H. Talimogene laherparepvec upregulates immune-cell populations in non-injected lesions: findings from a phase II, multicenter, open-label study in patients with stage IIIB-IVM1c melanoma. J Immunother Cancer. 2021 Mar;9(3):e001621. doi: 10.1136/jitc-2020-001621. PMID 33785610
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 36 centers across 12 countries in Europe from 07 April 2015 to 25 December 2020.
Period: Overall Study
Arm/Group | Talimogene Laherparepvec
Started | 112
Received Study Drug | 111
Completed | 58
Not Completed | 54
Not completed — Protocol-specified criteria | 3
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 1
Not completed — Death | 41

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of talimogene laherparepvec.
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 110
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 0
  Multiple | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 111
  Other | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active, no restrictions) | 87
    1 (Restricted but ambulatory) | 24
Log2(Intratumoral Cluster of Differentiation 8-positive (CD8+) Cell Density) [Mean (Standard Deviation); unit: Log2 CD8+ cells/mm²] — CD8+ cell density was assessed from tumor biopsy samples using CD8-specific immunohistochemistry. Population: Participants with non-missing data. Baseline data is available for 91 participants who had data available for analysis at the time of primary completion (26 June 2017). Baseline data is also presented for 93 participants who had data available at final analysis (25 December 2020).
  Log2 CD8+ cells/mm²
    Primary completion: number analyzed (Participants) | 91
    Primary completion | 8.041 (1.903)
    Final analysis: number analyzed (Participants) | 93
    Final analysis | 8.109 (1.940)

OUTCOME MEASURES:

1. Primary Outcome: Odds Ratio of Baseline Intratumoral CD8+ Cell Density and Objective Response Rate
Description: A univariate logistic regression model was performed to evaluate baseline log2(CD8+ cell density) as a predictor of objective response.
  Response was assessed according to the modified version of the World Health Organization (WHO) response criteria. Objective response rate (ORR) was defined as the percentage of participants with a complete response (CR) or partial response (PR) according to the modified WHO criteria.
  The unadjusted odds ratio of log2(baseline intratumoral CD8+ cell density) for objective response rate is reported.
Time Frame: Intratumoral CD8+ cell density: Baseline. Response: every 12 weeks until disease progression beyond 6 months of treatment or the start of new anticancer therapy; median time on follow-up at primary completion = 59 weeks (min 3 to max 116 weeks)
Population: Participants who received at least 1 dose of talimogene laherparepvec with non-missing baseline CD8+ cell density data. Data is available for 91 participants who had data available for analysis at the time of primary completion (26 June 2017).
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 91
ratio | 1.11 [0.87 to 1.42]
Statistical Analysis 1: Comparison: Talimogene Laherparepvec; Test type: Other; p = 0.387, Regression, Logistic

2. Secondary Outcome: Odds Ratio of Baseline Intratumoral CD8+ Cell Density and Durable Response Rate
Description: A univariate logistic regression model was performed to evaluate baseline log2(CD8+ cell density) as a predictor of durable response.
  Response was assessed according to the modified version of the World Health Organization (WHO) response criteria. Durable response rate (DRR) was defined as the percentage of participants with an objective response lasting continuously for 6 months and starting any time within 12 months of initiating therapy.
  The unadjusted odds ratio of log2(baseline intratumoral CD8+ cell density) for durable response rate is reported.
  Primary completion is defined as PC and final analysis is defined as FA.
Time Frame: Intratumoral CD8+ cell density: Baseline. Response: every 12 weeks until disease progression beyond 6 months of treatment or the start of new anticancer therapy; median time on follow-up: PC: 59 weeks (3 to 116 weeks); FA: 108 weeks (2.7 to 245.6)
Population: Participants who received at least 1 dose of talimogene laherparepvec with non-missing baseline CD8+ cell density data. Data is available for 91 participants who had data available for analysis at the time of primary completion (26 June 2017). Data is also presented for 93 participants who had data available at final analysis (25 December 2020).
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 93
ratio
  Primary completion: number analyzed (Participants) | 91
  Primary completion | 1.40 [0.99 to 1.97]
  Final analysis | 1.18 [0.91 to 1.53]
Statistical Analysis 1: Comparison: Talimogene Laherparepvec; Test type: Other — Primary completion data; p = 0.056, Regression, Logistic
Statistical Analysis 2: Comparison: Talimogene Laherparepvec; Test type: Other — Final analysis data; p = 0.222, Regression, Logistic

3. Secondary Outcome: Hazards Ratio of Baseline Intratumoral CD8+ Cell Density and Duration of Response
Description: A Cox proportional hazards regression model was performed to evaluate baseline log2(CD8+ cell density) as a predictor of duration of response.
  Response was assessed according to the modified version of the World Health Organization (WHO) response criteria. Duration of response (DOR) is defined as the longest individual period from entering an objective response (CR/PR) to the first documented evidence of the participant no longer meeting the criteria for being in the response (i.e. an overall response of either stable disease [SD] as compared with baseline or progressive disease [PD]).
  The unadjusted hazard ratio of log2(baseline intratumoral CD8+ cell density) for duration of response is reported.
Time Frame: Intratumoral CD8+ cell density: Baseline. Response: every 12 weeks until disease progression beyond 6 months of treatment or the start of new anticancer therapy; median time on follow-up: PC: 59 weeks (3 to 116 weeks); FA: 108 weeks (2.7 to 245.6 weeks)
Population: Participants who received at least 1 dose of talimogene laherparepvec with an objective response at the time of primary completion or final analysis, and with baseline CD8+ cell density data.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 29
ratio
  Primary completion: number analyzed (Participants) | 27
  Primary completion | 0.74 [0.39 to 1.37]
  Final analysis | 0.91 [0.63 to 1.30]
Statistical Analysis 1: Comparison: Talimogene Laherparepvec; Test type: Other — Primary completion data; p = 0.335, Cox proportional hazards
Statistical Analysis 2: Comparison: Talimogene Laherparepvec; Test type: Other — Final analysis data; p = 0.597, Cox proportional hazards

4. Secondary Outcome: Correlation Between Baseline Intratumoral CD8+ Cell Density and Changes in Tumor Burden
Description: Pearson's correlation coefficient (r) was estimated to assess the relationship between baseline log2(CD8+ cell density) and the maximum decrease in measurable tumor burden.
  Tumor burden is the sum of the products of the 2 largest perpendicular diameters (SPD) for all index lesions selected at baseline.
  The Pearson's correlation coefficient (r) of log2(baseline intratumoral CD8+ cell density) and the maximum decrease in tumor burden is reported.
  Primary completion is defined as PC and final analysis is defined as FA.
Time Frame: Intratumoral CD8+ cell density: Baseline; Tumor burden: First dose of study drug until primary completion date (26 June 2017) or end of follow-up; median time on follow-up: PC: 59 weeks (3 to 116 weeks); FA: 108 weeks (2.7 to 245.6 weeks)
Population: Participants who received at least 1 dose of talimogene laherparepvec with available tumor burden data at primary completion or final analysis, and baseline CD8+ cell density data.
Measure: Number (95% Confidence Interval); unit: Pearson's correlation coefficient
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 85
Pearson's correlation coefficient
  Primary completion: number analyzed (Participants) | 82
  Primary completion | 0.03 [-0.19 to 0.24]
  Final analysis | 0.01 [-0.20 to 0.23]
Statistical Analysis 1: Comparison: Talimogene Laherparepvec; Test type: Other — Primary completion; p = 0.82, Fisher's Z transformation
Statistical Analysis 2: Comparison: Talimogene Laherparepvec; Test type: Other — Final analysis data; p = 0.90, Fisher's Z transformation

5. Secondary Outcome: Odds Ratio of Change From Baseline Intratumoral CD8+ Cell Density and Objective Response Rate
Description: A univariate logistic regression model was performed to evaluate change from baseline to week 6 in log2(CD8+ cell density) in uninjected tumors as a predictor of objective response.
  Response was assessed according to the modified version of the World Health Organization (WHO) response criteria. Objective response rate (ORR) was defined as the percentage of participants with a complete response or partial response according to the modified WHO criteria.
  The unadjusted odds ratio of log2(change from baseline intratumoral CD8+ cell density) for objective response rate is reported.
  Intratumoral CD8+ Cell density has been shortened to "CD8+ cell density" in the time frame due to character limit. Primary completion is defined as PC and final analysis is defined as FA.
Time Frame: CD8+ cell density: Baseline & Week 6. Response: every 12 weeks until disease progression beyond 6 months of treatment or the start of new anticancer therapy; median time on follow-up: PC: 59 weeks (3 to 116 weeks); FA: 108 weeks (2.7 to 245.6 weeks)
Population: Participants who received at least 1 dose of talimogene laherparepvec with baseline and week 6 CD8+ cell density data for uninjected lesions. Data is available for 59 participants who had data available for analysis at the time of primary completion (26 June 2017). Data is also presented for 63 participants who had data available at final analysis (25 December 2020).
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 63
ratio
  Primary completion: number analyzed (Participants) | 59
  Primary completion | 0.94 [0.72 to 1.24]
  Final analysis | 0.98 [0.76 to 1.27]
Statistical Analysis 1: Comparison: Talimogene Laherparepvec; Test type: Other — Primary completion data; p = 0.660, Regression, Logistic
Statistical Analysis 2: Comparison: Talimogene Laherparepvec; Test type: Other — Final analysis data; p = 0.881, Regression, Logistic

6. Secondary Outcome: Odds Ratio of Change From Baseline in Intratumoral CD8+ Cell Density and Durable Response Rate
Description: A univariate logistic regression model was performed to evaluate change from baseline to week 6 in log2(CD8+ cell density) in uninjected lesions as a predictor of durable response.
  Response was assessed according to the modified version of the World Health Organization (WHO) response criteria. Durable response rate (DRR) was defined as the percentage of participants with an objective response lasting continuously for 6 months and starting any time within 12 months of initiating therapy.
  The unadjusted odds ratio of log2(change from baseline in intratumoral CD8+ cell density) for durable response rate is reported.
  Intratumoral CD8+ Cell density has been shortened to "CD8+ cell density" in the time frame due to character limit. Primary completion is defined as PC and final analysis is defined as FA.
Time Frame: as for outcome 5
Population: Participants who received at least 1 dose of talimogene laherparepvec with baseline and week 6 CD8+ cell density data in uninjected lesions. Data is available for 59 participants who had data available for analysis at the time of primary completion (26 June 2017). Data is also presented for 63 participants who had data available at final analysis (25 December 2020).
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 63
ratio
  Primary completion: number analyzed (Participants) | 59
  Primary completion | 0.99 [0.69 to 1.44]
  Final analysis | 0.93 [0.68 to 1.25]
Statistical Analysis 1: Comparison: Talimogene Laherparepvec; Test type: Other — Primary completion data; p = 0.974, Regression, Logistic
Statistical Analysis 2: Comparison: Talimogene Laherparepvec; Test type: Other — Final analysis data; p = 0.612, Regression, Logistic

7. Secondary Outcome: Hazard Ratio of Change From Baseline in Intratumoral CD8+ Cell Density and Duration of Response
Description: A Cox proportional hazards regression model was performed to evaluate change from baseline in log2(CD8+ cell density) as a predictor of duration of response.
  Response was assessed according to the modified version of the World Health Organization (WHO) response criteria. Duration of response (DOR) is defined as the longest individual period from entering an objective response (CR/PR) to the first documented evidence of the participant no longer meeting the criteria for being in the response (i.e. an overall response of either stable disease [SD] as compared with baseline or progressive disease [PD]).
  The unadjusted hazard ratio of log2(change from baseline intratumoral CD8+ cell density) for duration of response is reported.
  Intratumoral CD8+ Cell density has been shortened to "CD8+ cell density" in the time frame due to character limit. Primary completion is defined as PC and final analysis is defined as FA.
Time Frame: as for outcome 5
Population: Participants who received at least 1 dose of talimogene laherparepvec with an objective response at either primary completion or final analysis, and with baseline and week 6 CD8+ cell density data for uninjected lesions.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 18
ratio
  Primary completion: number analyzed (Participants) | 16
  Primary completion | 1.28 [0.47 to 3.47]
  Final analysis | 1.12 [0.74 to 1.69]
Statistical Analysis 1: Comparison: Talimogene Laherparepvec; Test type: Other — Primary completion data; p = 0.626, Cox proportional hazards
Statistical Analysis 2: Comparison: Talimogene Laherparepvec; Test type: Other — Final analysis data; p = 0.579, Cox proportional hazards

8. Secondary Outcome: Correlation Between Change From Baseline in Intratumoral CD8+ Cell Density and Changes in Tumor Burden
Description: Pearson's correlation coefficient (r) was estimated to assess the relationship between change from baseline in log2(CD8+ cell density) in uninjected lesions and the maximum decrease in measurable tumor burden.
  Tumor burden is the sum of the products of the 2 largest perpendicular diameters (SPD) for all index lesions selected at baseline.
  The Pearson's correlation coefficient (r) of log2(change from baseline intratumoral CD8+ cell density) and the maximum decrease in tumor burden is reported.
  Intratumoral CD8+ Cell density has been shortened to "CD8+ cell density" in the time frame due to character limit. Primary completion is defined as PC and final analysis is defined as FA.
Time Frame: as for outcome 5
Population: Participants who received at least 1 dose of talimogene laherparepvec with available tumor burden data at primary completion or final analysis, and baseline and week 6 CD8+ cell density data for uninjected lesions.
Measure: Number (95% Confidence Interval); unit: Pearson's correlation coefficient
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 60
Pearson's correlation coefficient
  Primary completion: number analyzed (Participants) | 56
  Primary completion | -0.18 [-0.42 to 0.09]
  Final analysis | -0.19 [-0.43 to 0.06]
Statistical Analysis 1: Comparison: Talimogene Laherparepvec; Test type: Other — Primary completion data; p = 0.18, Pearson's correlation coefficient
Statistical Analysis 2: Comparison: Talimogene Laherparepvec; Test type: Other — Final analysis data; p = 0.14, Pearson's correlation coefficient

9. Secondary Outcome: Objective Response Rate
Description: Objective Response rate is defined as the percentage of participants with either a CR or PR based on Modified WHO Response Criteria.
  CR: Complete disappearance of all index lesions, all non-index lesions, and any new tumors which might have appeared. Any residual cutaneous or subcutaneous index lesions must be documented by representative biopsy to not contain viable tumor.
  PR: Disappearance of all index lesions with persistence of one or more non-index tumor(s), or, 50% or greater reduction in the 2 largest perpendicular diameters (SPD) of all index lesions as compared to baseline, and disappearance or persistence of non-index lesions.
Time Frame: Response was assessed every 12 weeks until PD beyond 6 months of treatment or the start of new anticancer therapy; median time on follow-up at time of primary completion: 59 weeks (3 to 116 weeks); final analysis: 108 weeks (2.7 to 245.6 weeks)
Population: All participants who received at least 1 dose of talimogene laherparepvec.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 111
percentage of participants
  Primary completion | 27.0 [19.0 to 36.3]
  Final analysis | 28.8 [20.6 to 38.2]

10. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was defined as the longest individual period from entering an objective response (CR/PR) to the first documented evidence of the participant no longer meeting the criteria for objective response (i.e. an overall response of either stable disease [SD] as compared with baseline or progressive disease [PD]).
  SD: Neither sufficient tumor shrinkage of index lesion to qualify for response (PR or CR) nor sufficient tumor increase of index lesion to qualify for PD, with no increase in size of non-index lesions.
  PD: A > 25% increase in the sum of the SPD of all index tumors since baseline, or the unequivocal appearance of a new tumor since the last response assessment time point, or unequivocal progression of one or more non-index lesions.
  Participants last reported to be either a CR or PR were censored at that time point.
Time Frame: as for outcome 9
Population: Participants who received at least 1 dose of talimogene laherparepvec with an objective response at either primary completion (26 June 2017) or final analysis (25 December 2020).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 32
months
  Primary completion: number analyzed (Participants) | 30
  Primary completion | NA [11.5 to NA] — Not reached at time of analysis as most participants were still in response.
  Final analysis | NA [14.1 to NA] — Not reached at time of analysis as most participants were still in response.

11. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure (TTF) was calculated from first dosing until one or more of the following: (1) clinically relevant disease progression (PDr); (2) death from any cause; (3) non clinically relevant disease progression (PDn) associated with a requirement for alternative therapy as the reason for ending treatment or start of new anti-cancer therapy. Participants with no event were censored at their last evaluable tumor assessment.
Time Frame: From first dose of study drug until primary completion date of 26 June 2017, or end of follow-up; median time on follow-up at primary completion was 59 weeks (3 to 116 weeks); final analysis was 108 weeks (2.7 to 245.6 weeks)
Population: Participants who received at least 1 dose of talimogene laherparepvec.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 111
months
  Primary completion | 8.1 [5.4 to 10.9]
  Final analysis | 8.1 [5.4 to 11.0]

12. Secondary Outcome: Durable Response Rate
Description: Durable response rate (DRR) was defined as the percentage of participants with an objective response (CR or PR) based on modified WHO response criteria lasting continuously for 6 months and starting any time within 12 months of initiating therapy.
Time Frame: as for outcome 9
Population: Participants who received at least 1 dose of talimogene laherparepvec.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 111
percentage of participants
  Primary completion | 13.5 [7.8 to 21.3]
  Final analysis | 21.6 [14.4 to 30.4]

13. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from the date of first dose to the date of death from any cause.
  OS time was censored at the last date the participant was known to be alive when the confirmation of death is absent or unknown.
Time Frame: as for outcome 11
Population: Participants who received at least 1 dose of talimogene laherparepvec.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 111
months
  Primary completion | NA [NA to NA] — Median overall survival was not reached due to the low number of deaths.
  Final analysis | NA [34.9 to NA] — Median overall survival was not reached due to the low number of deaths.

14. Secondary Outcome: Change From Baseline in Tumor Burden
Description: Tumor burden is the sum of the products of the 2 largest perpendicular diameters (SPD) for all index lesions selected at baseline.
  Change from baseline in tumor burden was assessed in participants with an objective response.
Time Frame: Baseline and Day 1 of cycle 6, 12 , 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, 102, 108, 114, and 120. The first cycle was 21 days and all subsequent cycles were 14 days.
Population: Participants who received at least 1 dose of talimogene laherparepvec with an objective response (CR or PR)
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 32
cm²
  Baseline | 16.420 (41.269)
  Change from baseline at Cycle 6 day 1 | -5.883 (12.158)
  Change from baseline at Cycle 12 day 1: number analyzed (Participants) | 30
  Change from baseline at Cycle 12 day 1 | -10.085 (22.862)
  Change from baseline at Cycle 18 day 1: number analyzed (Participants) | 23
  Change from baseline at Cycle 18 day 1 | -13.074 (27.798)
  Change from baseline at Cycle 24 day 1: number analyzed (Participants) | 15
  Change from baseline at Cycle 24 day 1 | -21.407 (42.221)
  Change from baseline at Cycle 30 day 1: number analyzed (Participants) | 12
  Change from baseline at Cycle 30 day 1 | -30.404 (55.593)
  Change from baseline at Cycle 36 day 1: number analyzed (Participants) | 10
  Change from baseline at Cycle 36 day 1 | -31.803 (69.358)
  Change from baseline at Cycle 42 day 1: number analyzed (Participants) | 9
  Change from baseline at Cycle 42 day 1 | -10.208 (14.188)
  Change from baseline at Cycle 48 day 1: number analyzed (Participants) | 8
  Change from baseline at Cycle 48 day 1 | -11.396 (14.885)
  Change from baseline at Cycle 54 day 1: number analyzed (Participants) | 8
  Change from baseline at Cycle 54 day 1 | -11.693 (15.720)
  Change from baseline at Cycle 60 day 1: number analyzed (Participants) | 6
  Change from baseline at Cycle 60 day 1 | -13.122 (17.791)
  Change from baseline at Cycle 66 day 1: number analyzed (Participants) | 6
  Change from baseline at Cycle 66 day 1 | -16.797 (14.659)
  Change from baseline at Cycle 72 day 1: number analyzed (Participants) | 6
  Change from baseline at Cycle 72 day 1 | -16.797 (14.659)
  Change from baseline at Cycle 78 day 1: number analyzed (Participants) | 6
  Change from baseline at Cycle 78 day 1 | -16.858 (14.730)
  Change from baseline at Cycle 84 day 1: number analyzed (Participants) | 6
  Change from baseline at Cycle 84 day 1 | -17.022 (14.992)
  Change from baseline at Cycle 90 day 1: number analyzed (Participants) | 5
  Change from baseline at Cycle 90 day 1 | -13.916 (14.381)
  Change from baseline at Cycle 96 day 1: number analyzed (Participants) | 4
  Change from baseline at Cycle 96 day 1 | -16.505 (15.244)
  Change from baseline at Cycle 102 day 1: number analyzed (Participants) | 3
  Change from baseline at Cycle 102 day 1 | -17.793 (18.413)
  Change from baseline at Cycle 108 day 1: number analyzed (Participants) | 3
  Change from baseline at Cycle 108 day 1 | -17.733 (18.426)
  Change from baseline at Cycle 114 day 1: number analyzed (Participants) | 1
  Change from baseline at Cycle 114 day 1 | -1.694 (NA) — Only 1 participant had non-missing data at this time-point, so standard deviation could not be calculated.
  Change from baseline at Cycle 120 day 1: number analyzed (Participants) | 1
  Change from baseline at Cycle 120 day 1 | -39.930 (NA) — Only 1 participant had non-missing data at this time-point, so standard deviation could not be calculated.

15. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity of each adverse event (AE) was assessed according to the Common Terminology Criteria for Adverse Events (CTCAE), version 3.0 grading scale, where Grade 1 = Mild AE Grade 2 = Moderate AE Grade 3 = Severe AE Grade 4 = Life-threatening or disabling AE Grade 5 = Death related to AE Treatment-related adverse events (TRAE) were those assessed by the investigator as possibly related to talimogene laherparepvec.
Time Frame: From first dose through 30 days after last dose of talimogene laherparepvec; median duration of treatment was 25.143 weeks (range 0.14 to 241.43 weeks)
Population: Participants who received at least 1 dose of talimogene laherparepvec.
Measure: Count of Participants; unit: Participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 111
Participants
  Any adverse event | 108
  Adverse events ≥ grade 3 | 38
  Adverse events ≥ grade 4 | 11
  Serious adverse events | 33
  AE leading to discontinuation of study drug | 4
  Fatal adverse events | 4
  Treatment-related adverse events | 93
  Treatment-related adverse events ≥ grade 3 | 11
  Treatment-related adverse events ≥ grade 4 | 2
  Treatment-related serious adverse events | 9
  TRAE leading to discontinuation of study drug | 3
  Treatment-related fatal adverse events | 0

ADVERSE EVENTS:
Time Frame: Deaths are reported from enrollment through to end of follow-up; median time on follow up was 108 weeks (2.7 to 245.6 weeks). Adverse events are reported from first dose through 30 days after last dose of talimogene laherparepvec; median duration of treatment was 25.143 (0.14 to 241.43 weeks)
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Talimogene Laherparepvec
All-Cause Mortality (participants affected / at risk) | 41/112
Serious Adverse Events (participants affected / at risk) | 33/111
Other Adverse Events (participants affected / at risk) | 97/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec (N=111)
Cardiac failure (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 2
Pyrexia (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Medical observation (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anxiety (Psychiatric disorders) | 1
Paranoia (Psychiatric disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Oedema peripheral (General disorders) | 1
Neurofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardiac pacemaker replacement (Surgical and medical procedures) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Ileus (Gastrointestinal disorders) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec (N=111)
Abdominal pain (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 26
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 18
Chills (General disorders) | 30
Fatigue (General disorders) | 24
Influenza like illness (General disorders) | 29
Injection site pain (General disorders) | 19
Pain (General disorders) | 7
Pyrexia (General disorders) | 52
Decreased appetite (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 20
Back pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Headache (Nervous system disorders) | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Oedema peripheral (General disorders) | 7
Nasopharyngitis (Infections and infestations) | 11
Anaemia (Blood and lymphatic system disorders) | 8
Erythema (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT02366195/Prot_000.pdf
  • Statistical Analysis Plan (2014-08-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT02366195/SAP_001.pdf